CLINICAL TRIAL: NCT01581892
Title: Treatment of Long Bone Nonunion With Autologous Bone Marrow Stem Cells. Phase I/II Study
Brief Title: Use of Adult Bone Marrow Mononuclear Cells in Patients With Long Bone Nonunion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Central de Asturias (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUCA
Record Dates: First submitted 2012-04-09; First posted 2012-04-20 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Long Bone Nonunion
Keywords: bone nonunion; bone marrow; mononuclear; fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Fracture Fixation, Internal; leukocyte procoagulant activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone marrow stem cells (Experimental): Bone marrow is obtained by posterosuperior iliac crest aspiration under topical anesthesia. Mononuclear cells were isolated by Ficoll density gradient and will be resuspended in heparinized isotonic saline for mixing with osteogenic matrix.
  Interventions: Procedure: Osteosynthesis

INTERVENTIONS:
Procedure: Osteosynthesis — To mix the cell suspension with osteogenic matrix and to use sheet and nails in order to consolidate the fracture
  Other Names: bone nonunion; bone marrow; mononuclear; fracture

SUMMARY:
The aim of the study is to determine the safety and feasibility of autologous mononuclear stem cells in long bone nonunion; and moreover, to evaluate the efficacy of the treatment.

DETAILED DESCRIPTION:
In this study the investigators examine the improvement of conventional surgical treatment of long bone nonunion with the administration of bone marrow stem cells in order to achieve a higher percentage of healing and tissue reparation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed long bone nonunion
* age from 18 years old

Exclusion Criteria:

* active infection
* cancer patients
* concomitant serious illness
* pregnant women
* evidences of mental illness
* previous alcohol or drug dependences
* previous malignant disease during last 5 years, except for basal carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Absence of adverse effects during timeframe as infections or complications related with the intervention | Six months
  The proposed trial will involve the recruitment of a total of 30 patients. The cells will be collected via bone marrow sampling. The aspirate will be centrifuged on a Ficoll density gradient to isolate mononuclear cells, wich will be resuspended in heparinized isotonic saline and used in order to infuse into the area surgically treated. The surgical intervention means the introduction of a sheet with nails according with the usually employed technique.

SECONDARY OUTCOMES:
Improvement and union of the bone | One year
  The improvement of the bone nonunion will be assessed by X-ray and NMR

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Otero, MD, Principal Investigator — Unidad de Coordinación de Trasplantes, Terapia Celular y Medicina Regenerativa
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

REFERENCES:
- [Background] Fernandez-Bances I, Perez-Basterrechea M, Perez-Lopez S, Nunez Batalla D, Fernandez Rodriguez MA, Alvarez-Viejo M, Ferrero-Gutierrez A, Menendez-Menendez Y, Garcia-Gala JM, Escudero D, Paz Aparicio J, Carnero Lopez S, Lopez Fernandez P, Gonzalez Suarez D, Otero Hernandez J. Repair of long-bone pseudoarthrosis with autologous bone marrow mononuclear cells combined with allogenic bone graft. Cytotherapy. 2013 May;15(5):571-7. doi: 10.1016/j.jcyt.2013.01.004. Epub 2013 Feb 14. PMID 23415918